CLINICAL TRIAL: NCT02244372
Title: A 8-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Cordyceps Sinensis Mycelium Culture Extract(Paecilomyces Hepiali, CBG-CS-2) on Promotion of Immunity
Brief Title: Efficacy and Safety of Cordyceps Sinensis Mycelium Culture Extract(Paecilomyces Hepiali, CBG-CS-2) on Promotion of Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHE-PI-CM
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Immunity
Keywords: Cordyceps sinensis mycelium culture extract(Paecilomyces hepiali, CBG-CS-2); immunity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cordyceps sinensis mycelium culture extract 0.76 g (Experimental): Cordyceps sinensis mycelium culture extract 0.76 g
  Interventions: Dietary Supplement: Cordyceps sinensis mycelium culture extract 0.76 g
- Cordyceps sinensis mycelium culture extract 1.15 g (Experimental): Cordyceps sinensis mycelium culture extract 1.15 g
  Interventions: Dietary Supplement: Cordyceps sinensis mycelium culture extract 1.15 g
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cordyceps sinensis mycelium culture extract 0.76 g
  Arms: Cordyceps sinensis mycelium culture extract 0.76 g
Dietary Supplement: Cordyceps sinensis mycelium culture extract 1.15 g
  Arms: Cordyceps sinensis mycelium culture extract 1.15 g
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The investigators performed randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Cordyceps sinensis mycelium culture extract (Paecilomyces hepiali, CBG-CS-2) on promotion of immunity. The investigators measured promotion of immunity parameters , including Cytotoxicity, Cytokine (IL-4, IL-6, IL-12, IFN-γ, TNF-α), hs-CRP, antibody titer, and upper respiratory tract infection(URI)

ELIGIBILITY:
Inclusion Criteria:

* Males and females 20-80 years old
* Who had suffered more than twice Upper respiratory infection* disorder or common cold causing URI
* Able to give informed consent

Exclusion Criteria:

* WBC concentration below 3000 ㎕
* Subjects vaccinated against influenza within the last 6 months prior to the study
* Subjects with Upper respiratory infection at screening visit
* Subjects with BMI < 18.5 kg/m2 at screening visit
* Allergic or hypersensitive to any of the ingredients in the test products
* Diagnosed of gastrointestinal disease such as Immune-related diseases, severe hepatic, renal failure, and diabetes
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in Cytotoxicity | 4, 8 weeks
  Cytotoxicity was measured in study visit 1(0 week), visit 2(4 week) and visit 3(8 week). cytotoxicity was measured by NK cell activity.
  Cytotoxicity (%) = (experimental release - spontaneous release) / (maximum release - spontaneous release) x 100

SECONDARY OUTCOMES:
Changes in Cytokine(IL-4, IL-6, IL-12, IFN-γ, TNF-α) | 4, 8 weeks
  Cytokine(IL-4, IL-6, IL-12, IFN-γ, TNF-α) was measured in study visit 1(0 week), visit 2(4 week), and visit 3(8 week).
Changes in hs-CRP | 4, 8 weeks
  hs-CRP was measured in study visit 1(0 week), visit 2(4 week) and visit 3(8 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea